CLINICAL TRIAL: NCT06944327
Title: Reduction of Complications Associated With PICC Management. Randomization in Care.
Brief Title: Reduction of Complications Associated With PICC Management
Acronym: PICC managemen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Complejo Hospitalario de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Quality_PICC; Quality_PICC (Other: Fundacion Miguel Servet)
Record Dates: First submitted 2025-04-03; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Treatment Outcome; Vascular Access; Vascular Access Device; Vascular Access Complication; Care Delivery; Nurse; Nurse Based Care Management
Keywords: vascular; vascular access; catheter; central catheter; nurse; vascular access device; management; complication

STUDY DESIGN:
Intervention Model Description: Randomized prospective longitudinal design, by means of a representative sample selection of the study population, in a simple randomized fashion.
  The study will be conducted and piloted at the Hospital Universitario de Navarra, in the Intravenous Therapy Unit (ITU).
  A certain number of patients who meet the inclusion criteria (representative sample of the population to be studied) will be registered and analyzed during the same period (6 months) to determine and record the study variables and outcome data.
  In this case, the inclusion criteria for taking part in the study will be all patients over 18 years of age, with a level of independence for optimal care and attended in the ICU for the insertion of a long-term PIVC device who voluntarily accept to participate in the study.
  As selection criteria, all cases of dependent, bedridden and hemodynamically unstable patients will be considered as exclusion criteria, as well as all users who, after informing the patients or legal guardians
Who Masked: Participant, Investigator
Masking Description: To conduct effective masking in a quasi-experimental study of catheter care, it is critical to implement a design that minimizes bias for both patients and investigators. First, patients should be randomly assigned to different intervention groups, ensuring that they have no knowledge about the type of care they will receive (e.g., standard care versus a new care protocol). This can be accomplished through the use of sealed envelopes or an online allocation system that keeps randomization hidden. On the other hand, investigators assessing outcomes should also be masked to patient assignment; this can be achieved by forming an independent team to perform the assessments and data analysis, without access to information about which group each patient belongs to. In addition, training should be provided to all personnel involved in the study to ensure that blinding procedures are followed and the integrity of the study is maintained. In this way, biases are minimized and the validity of th
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PIVC fixed with SecurAcath 7 DAYS (Placebo Comparator): G1: PIVC fixed with SecurAcath, with care performed by heparinization with push-stop-push technique and positive pressure + fibrillin and semitransparent dressing change (Tergaderm 3M fully reinforced membrane dressing (TSM) every 7 days.
  Interventions: Other: traditional care
- PIVC fixed with SecurAcath 14 DAYS (Experimental): G2: PIVC fixed with SecurAcath, with care performed by heparinization with push-stop-push technique and positive pressure + fibrillin and dressing change dressing 7 semitransparent (fully reinforced membrane dressing (TSM) Tergaderm 3M every 14 days.
  Interventions: Procedure: MANAGEMENT CARE
- PIVC fixed with SecurAcath with Derma+ Flex® QS Skin Tissue Adhesive 7 days (Experimental): G3: PIVC fixed with SecurAcath PLUS Derma+ Flex® QS Skin Tissue Adhesive, with care performed by heparinization with push-stop-push technique and positive pressure + sealing solution + saline and semitransparent dressing change (Tergaderm 3M fully reinforced membrane dressing (TSM) every 7 days.
  Interventions: Procedure: MANAGEMENT CARE
- SecurAcath + Derma+ Flex® QS Skin Tissue Adhesive14 days (Experimental): PIVC fixed with SecurAcath PLUS Derma+ Flex® QS Skin Tissue Adhesive, with care performed by heparinization with push-stop-push technique and positive pressure + saline + sealing solution+ saline and semitransparent dressing change (Tergaderm 3M fully reinforced membrane dressing (TSM) every 14 days.
  Interventions: Procedure: MANAGEMENT CARE

INTERVENTIONS:
Procedure: MANAGEMENT CARE — Administration of the sealing element after canalization and initial treatment of the device, prior to fixation with a suture system and a 7-day vs. 14-day cadence test.
  Arms: PIVC fixed with SecurAcath 14 DAYS; PIVC fixed with SecurAcath with Derma+ Flex® QS Skin Tissue Adhesive 7 days; SecurAcath + Derma+ Flex® QS Skin Tissue Adhesive14 days
Other: traditional care — Traditional cure administration with sutureless device fixation every 7 days
  Arms: PIVC fixed with SecurAcath 7 DAYS

SUMMARY:
The present study aims to analyze different care routes of the peripheral access central venous catheter to assess which alternative allows a moderate reduction in the level of complications associated with prolonged care frequency, due to the reduction of device manipulation.

A high level of patient satisfaction is detected due to the controlled follow-up of the device care, as well as a decrease in the need for transfer to a center for follow-up.

Objective: Identify the type of care frequency for PIVCs most beneficial for the reduction of complications associated with extraluminal device care (thrombosis, phlebitis, accidental removal, obstruction).

DETAILED DESCRIPTION:
Study variables and measurement instruments:

Sociodemographic and control variables: age and sex, reason for admission, clinical diagnosis, day of care.

Device-related variables: Catheter type, brand, access type, caliber, number of lumens, infusion/pharmacological therapy, number of simultaneous therapies, days of access cannulation, frequency of care, antiseptic used in access manipulation, dressing and fixation system, other device care, direct and indirect costs.

Dependent variables: Complications (infectious, mechanical, chemical, or thrombotic), reason for removal and accidental dislodgement, cost, patient satisfaction level.

Data collection:

The catheter will be inserted by the Intravenous Therapy Unit, which will provide the patient with information and sign a consent form prior to participation in the study. After the insertion process, the device placement representative will record the device characteristics and relevant aspects of the insertion, generating a 1-1 random assignment of the study participation group.

This assignment will be done by giving the patient a code during the data entry process. This will allow for blinding of subsequent data collection and proper, anonymous follow-up of the case.

Once insertion is complete, the device will be secured by applying Dermabond Mini glue (2-Octyl Cyanoacrylate), the SecurAcath system (a subcutaneous stabilization device that does not require changing while the catheter is in place), and a semi-transparent dressing (3M Tergaderm fully reinforced membrane (TSM) dressing), which will allow for monitoring the insertion site and randomizing care.

Once the study group has been assigned and the device has been placed, patient follow-up, including standardized device treatment at 7 days, will be conducted by a trained professional dedicated exclusively to this care. Follow-up data will be collected: date of treatment, treatment and elements used, and findings on the device or patient. The follow-up process will be blinded at all times by both the professional and the patient.

After the established 6-month follow-up period, a patient satisfaction questionnaire will be completed, and the coded data will be reported for assessment and interpretation by the research team.

Likewise, an analysis of the economic costs involved in each care frequency will be performed, thanks to the collaboration of the center's financial management service, which will calculate the average direct and indirect costs resulting from each care frequency.

Data Analysis:

The collected data will be pre-coded by the research team, ensuring the anonymity of the data and all participants. The results will be recorded in the SPSS statistical software so that they can be analyzed and processed directly. For analysis and interpretation, support is provided by statistical experts within the research group, as well as by an institution that collaborates with some team members.

Ethical Aspects:

A request from the Research Ethics Committee has been made. Likewise, information for participants and family members is ensured through a written report that includes a comprehensive explanation of the project and participant rights. This report will be delivered after verbal communication and any questions are resolved. After verbal acceptance of participation in the process, a paper informed consent form is provided for the patient or legal guardian to sign.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years of age
* accept participation in the study
* independent patient in the care and management of activities of daily living

Exclusion Criteria:

* patient over 18 years of age
* patient with functional or cognitive limitation
* patient with mild, moderate or high level of dependence
* patient does not accept to perform the study
* patient with device withdrawal prior to 14 days of duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify the type of frequency of care for PIVCs most beneficial for the reduction of complications associated with extraluminal device care (LESS thrombosis, phlebitis, accidental removal, obstruction). | Measurement follow-up until removal or 6 and 12 months after catheter implantation.
  Reduction of complications such as thrombosis, phlebitis, accidental withdrawals, obstruction. measurement of the various complications according to: number of associated complications per device according to intervention group

SECONDARY OUTCOMES:
level of patient satisfaction related to various processes and frequencies of care | day 1, day 7, day 14, at 6 months after placement and start of the study of the device and at 12 months after the device is removed.
  use of a liker-type scale to determine the level of overall satisfaction with the care and handling of the device

OTHER OUTCOMES:
Recognize the cost-effectiveness of each of the randomization groups included in the study. | day 1, day 7, day 14, at 6 months after placement and start of the study of the device and at 12 months after the device is removed. at 6 months after placement and start of the study of the device and at 12 months after the device is removed
  Measurement of direct and indirect costs of device care by study group, taking into account whether there are complications and the costs associated with them.

IPD SHARING:
Plan to Share IPD: No